CLINICAL TRIAL: NCT03290469
Title: NICUSeq: A Prospective Trial to Evaluate the Clinical Utility of Human Whole Genome Sequencing (WGS) Compared to Standard of Care in Acute Care Neonates and Infants
Brief Title: NICUSeq: A Trial to Evaluate the Clinical Utility of Human Whole Genome Sequencing (WGS) Compared to Standard of Care in Acute Care Neonates and Infants
Acronym: NICU-Seq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illumina, Inc. (Industry)
Collaborators: Le Bonheur Children's Hospital (Other); Rady Pediatric Genomics & Systems Medicine Institute (Other); Children's Hospital of Orange County (Other); Children's Hospital and Medical Center, Omaha, Nebraska (Other); St. Louis Children's Hospital (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NICU-R001
Record Dates: First submitted 2017-09-13; First posted 2017-09-25 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2019-05

CONDITIONS: Rare Diseases
Keywords: ICU; Intensive Care Unit
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Intervention Model Description: Multi-cohort, time delay study receiving Clinical Whole Genome Sequencing (cWGS) at either 15 days or 60 days in an acutely ill newborn population
Who Masked: Participant, Care Provider, Investigator
Masking Description: All investigators are masked to the study arm until Day 15 to ensure SOC throughout first 15 days on study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 day cWGS and Standard of Care (Experimental): Enrolled cohorts receive the results of the clinical whole genome sequencing (cWGS) after 15 days of the sample receipt while still undergoing standard of care (SOC).
  Interventions: Other: clinical whole genome sequencing (cWGS)
- Standard of Care (No Intervention): Enrolled cohorts receive the results of the clinical whole genome sequencing (cWGS) after 60 days of the sample receipt while still undergoing standard of care (SOC).

INTERVENTIONS:
Other: clinical whole genome sequencing (cWGS) — Clinical Whole Genome Sequencing (cWGS) consists of the sequencing, analysis and interpretation of subjects samples and a return of the result to the ordering physician.
  Arms: 15 day cWGS and Standard of Care

SUMMARY:
Prospective, multi-site, study to evaluate the clinical utility of cWGS in a proband. One group will receive cWGS and a clinical report approximately 15 days after blood samples are received, while the other group will continue to receive standard of care until Day 60. The standard of care group will receive cWGS and a clinical report at Day 60 as part of secondary and tertiary analyses. Both groups will be followed for a total of 90 days.

DETAILED DESCRIPTION:
This is a prospective, multi-site, randomized study to evaluate the clinical utility of cWGS in each proband. Throughout this study, each proband will receive SOC testing as determined by the site clinical team. Upon enrollment in the study, each proband will be randomly assigned to the 15 day cWGS group or the SOC group. SOC is defined as the management of the proband's care under the same or similar conditions as if the proband was not enrolled in this study. A blood sample from each enrolled proband will be collected and shipped to the Illumina Clinical Services Laboratory ("ICSL"), which is Clinical Laboratory Improvement Amendments (CLIA)-certified and College of American Pathologists (CAP)-accredited. ICSL will conduct cWGS testing with the TruGenome Undiagnosed Disease Test ("TruGenome Test"). The TruGenome Test cWGS results will be provided to the Principal Investigator (PI) or designee who will evaluate each proband test outcome based on the aggregate medical information, informed by the cWGS or SOC results.

ELIGIBILITY:
Proband Inclusion Criteria

1. Current admission in a Neonatal Intensive Care Unit/Intensive Care Unit at a participating clinical site at the time of enrollment from day of life 0 to 120 days
2. A suspected genetic etiology of disease, based on objective clinical findings or other phenotypic defects for which a genetic test would be considered
3. Must be able to have 1 - 1.25 ml tube of whole blood drawn for testing
4. One parent of the proband must be able to provide written informed consent
5. At least one biological parent must agree to participate and provide at least 4 ml of whole blood for testing

Exclusion Criteria:

Proband Exclusion Criteria

1. Known non-genetic cause(s) of disease, disorder, or phenotypic defect
2. The phenotype is fully explained by complications of prematurity
3. Trisomy 13, 18 or 21 or Turner Syndrome is the likely diagnosis; such a proband will be eligible if a diagnostic karyotype is normal
4. Blood transfusion within 48 hours (each proband will be re-eligible 48 hours after the most recent transfusion)
5. The PI decides that the study is not in the best interest of the proband (for example, the neonate or infant is at a high risk of severe morbidity or mortality within the next 7 days and these risks could be mitigated by alternative testing). Subsequent eligibility for enrollment of each proband is at the discretion of the site PI.

Ages: 1 Day to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 355 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
A difference in Change of Management between the 15 day cWGS and standard of care groups | Day 60
  Change of Management is a binary (yes or no) based on assignments made by the PI or designee at each site using the following domains:
  * Condition specific management
  * Condition specific supportive interventions
  * Palliative care/End of Life Care A change in any of these domains will be considered a change of management.

SECONDARY OUTCOMES:
Diagnostic Yield | 90 Days
  Diagnostic yield (# positive diagnoses/ total # of each proband expressed as a percentage)
Diagnostic Accuracy | 90 Days
  Diagnostic accuracy (percent positive agreement between test outcome classified by the medical monitor and the site PI or designee)
  % diagnoses returned before discharge or death
Genetic Results Returned | 90 Days
  % diagnoses returned before discharge or death
Costs | 90 Days
  Pre-test costs of hospital care
Average Time to Diagnosis | 90 Days
  Average time (in days) to diagnose between cWGS and SOC based on the comparison of the (a) cWGS results and the (b) current clinical diagnoses
The amount of imaging tests ordered as assessed by counting the number of tests per cohort. | 90 Days
  Clinical services utilization includes the number of imaging tests ordered.
cWGS satisfaction questionnaire will be given to clinicians and families at the conclusion of the study. | 90 Days
  The questionnaire is a likard scale questionnaire developed by the study team to assess satisfaction levels from the perspective of the clinician and also the parent.
Assessment of Clinical Utility by using a questionnaire | 90 Days
  A questionnaire developed by the study team will assess the Clinical Utility of the cWGS test
Change in Care Setting from the ICU environment | 90 Days
  Changes in care level setting from the ICU environment will be compared between the 15 day cWGS group and the SOC group.
Time to diagnosis | 90 Days
  Time to diagnosis (in days of life)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J. Taft, PhD, Study Director — Illumina, Inc.
Locations (5):
- United States (5):
  - Rady's/Children's Hospital of Orange County, Orange, California
  - Washington University in St. Louis School of Medicine & St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center & Children's Hospital, Omaha, Nebraska
  - Children's Hospital of Philadelpia, Philadelphia, Pennsylvania
  - LeBonheur Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
Deidentified and curated variant and limited phenotype information will be submitted to ClinVar. ClinVar is a freely accessible, public archive of reports of the relationships among human variations and phenotypes hosted by the National Center for Biotechnology Information (NCBI) and funded by Intramural National Institutes of Health (NIH) funding. No personal health information (PHI) or information identifying the participant or family will be submitted.

REFERENCES:
- [Derived] NICUSeq Study Group; Krantz ID, Medne L, Weatherly JM, Wild KT, Biswas S, Devkota B, Hartman T, Brunelli L, Fishler KP, Abdul-Rahman O, Euteneuer JC, Hoover D, Dimmock D, Cleary J, Farnaes L, Knight J, Schwarz AJ, Vargas-Shiraishi OM, Wigby K, Zadeh N, Shinawi M, Wambach JA, Baldridge D, Cole FS, Wegner DJ, Urraca N, Holtrop S, Mostafavi R, Mroczkowski HJ, Pivnick EK, Ward JC, Talati A, Brown CW, Belmont JW, Ortega JL, Robinson KD, Brocklehurst WT, Perry DL, Ajay SS, Hagelstrom RT, Bennett M, Rajan V, Taft RJ. Effect of Whole-Genome Sequencing on the Clinical Management of Acutely Ill Infants With Suspected Genetic Disease: A Randomized Clinical Trial. JAMA Pediatr. 2021 Dec 1;175(12):1218-1226. doi: 10.1001/jamapediatrics.2021.3496. PMID 34570182